CLINICAL TRIAL: NCT01304524
Title: Phase II Placebo Controlled Study of VGX-3100, (HPV16 E6/E7, HPV18 E6/E7 DNA Vaccine) Delivered IM Followed by Electroporation With CELLECTRA-5P for the Treatment of Biopsy-proven CIN 2/3 or CIN 3 With Documented HPV 16 or 18.
Brief Title: A Study of VGX-3100 DNA Vaccine With Electroporation in Patients With Cervical Intraepithelial Neoplasia Grade 2/3 or 3
Acronym: HPV-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPV-003
Record Dates: First submitted 2011-02-16; First posted 2011-02-25 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: CIN 2/3 or CIN 3; Cervical cancer; Papillomavirus
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- VGX 3100 (Experimental)
  Interventions: Biological: VGX 3100; Device: CELLECTRA™-5P
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo; Device: CELLECTRA™-5P

INTERVENTIONS:
Biological: VGX 3100 — 1ml of VGX-3100 delivered IM followed by electroporation at Day 0, Week 4 and Week 12.
  Arms: VGX 3100
Biological: Placebo — 1ml of placebo delivered IM followed by electroporation at Day 0, Week 4 and Week 12.
  Arms: Placebo
Device: CELLECTRA™-5P — CELLECTRA™-5P is used for electroporation following IM delivery of VGX 3100 or placebo on Day 0, Week 4 and Week 12.

SUMMARY:
This is randomized, placebo controlled study to determine safety and efficacy of VGX-3100 DNA Vaccine delivered by Electroporation to adult women with biopsy-proven HPV 16 or 18 associated Cervical intraepithelial neoplasia grade 2/3 or 3.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects age 18-55 years;
* Histologically confirmed HPV-16 or HPV-18-associated CIN 2/3 or CIN 3 from tissue collected less than 10 weeks prior to Vaccination/EP #1 with no evidence of invasive cancer in any specimen;
* Colposcopy is satisfactory based on visualization of the entire squamocolumnar junction and the upper limit of the entire aceto-white or suspected CIN disease area; lesions in ≤ 3 cervical quadrants (4 quadrant disease where the lesion occupies less than 50% of each quadrant will be considered for inclusion);
* Healthy subjects as judged by the Investigator based on medical history, PE, and normal results for an ECG, CBC, Serum Chemistries, CPK and urinalysis done up to 4 weeks prior to enrollment and administration of study drug;
* Women of child-bearing potential agree to remain sexually abstinent, use two medically effective methods of contraception (e.g. oral contraception, barrier methods, spermicide, intrauterine device (IUD)), or have a partner who is sterile (i.e., vasectomy) through 36 weeks (9 months);
* Able and willing to comply with all study procedures and voluntarily signs informed consent form

Exclusion Criteria:

* Unsatisfactory colposcopy defined as incomplete visualization of the entire squamocolumnar junction and the upper limit of the entire aceto-white or suspected CIN disease area;
* Pregnancy or breastfeeding
* Immunosuppression including any concurrent condition requiring the continued use of systemic or topical steroids at or near the injection site [deltoid, upper arm] (excluding inhaled and eye drop-containing corticosteroids) or the use of immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 0 of study vaccine administration; autoimmune disorders, transplant recipients;
* History of previous therapeutic HPV vaccination (individuals who have been immunized with licensed prophylactic HPV vaccines (e.g. Gardasil®, Cervarix®) are not excluded);
* Positive serological test for hepatitis C virus or hepatitis B virus surface antigen(HBsAg) or human immunodeficiency virus (HIV)
* Administration of any blood product within 3 months of enrollment
* Administration of any licensed vaccine within 2 weeks of enrollment( 4weeks for measles vaccine)
* Participation in a study with an investigational compound or device within 30 days of signing informed consent;
* Cardiac pre-excitation syndromes (such as Wolff-Parkinson-White);
* History of seizures (unless seizure free for 5 years);
* Tattoos, scars, or active lesions/rashes within 2 cm of the intended site of vaccination/EP or any implantable leads; or any implantable leads;
* Active drug or alcohol use or dependence that, in the opinion of the investigator,would interfere with adherence to study requirements;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated)for treatment of either a psychiatric or physical (i.e. infections disease) illness must not be enrolled into this study;
* Any other conditions judged by the investigator that would limit the evaluation of a subject

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2011-04; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Histopathological Regression of Cervical Lesions to CIN 1 or Less as a Measure of Efficacy. | 36 weeks
  The number of participants with histopathologically confirmed CIN2/3 or CIN 3 associated with HPV16 or HPV18 whose cervical lesions regress to CIN 1 or less at the 36 week visit.

SECONDARY OUTCOMES:
Number of Participants with Virologically-proven Clearance of HPV 16 or 18 in Combination with Histopathological Regression of Cervical Lesions to CIN 1 or Less as a Secondary Measure of Efficacy | 36 Weeks
  The number of participants with histopathologically confirmed CIN2/3 or CIN 3 associated with HPV16 or HPV18 whose cervical lesions regress to CIN 1 or less and have virologically-proven clearance of HPV16 or HPV18 at the 36 week visit.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Trimble, MD, Principal Investigator — Johns Hopkins University; Robert L Parker, Jr., MD, Principal Investigator — Lyndhurst Gynecologic Associates
Locations (43):
- United States (27):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Colton, California
  - La Mesa, California
  - Los Angeles, California
  - Lakewood, Colorado
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Sarasota, Florida
  - Baltimore, Maryland
  - Saginaw, Michigan
  - Missoula, Montana
  - Port Jefferson, New York
  - The Bronx, New York
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Philadelphia, Pennsylvania
  - Myrtle Beach, South Carolina
  - Murray, Utah
  - Pleasant Grove, Utah
  - Sandy City, Utah
  - Richmond, Virginia
  - Renton, Washington
  - Spokane, Washington
- Victoria, Australia
- Canada (2):
  - Montreal, Quebec
  - Vancouver
- Estonia (2):
  - Tallinn
  - Tartu
- Georgia (2):
  - Batumi
  - Tbilisi
- India (5):
  - Bangalore, Karnataka
  - Jaipur, Rajasthan
  - Kolkata
  - New Delhi
  - Pune
- San Juan, Puerto Rico
- South Africa (2):
  - Bloemfontein
  - Cape Town
- Seoul, South Korea

REFERENCES:
- [Derived] Bhuyan PK, Dallas M, Kraynyak K, Herring T, Morrow M, Boyer J, Duff S, Kim J, Weiner DB. Durability of response to VGX-3100 treatment of HPV16/18 positive cervical HSIL. Hum Vaccin Immunother. 2021 May 4;17(5):1288-1293. doi: 10.1080/21645515.2020.1823778. Epub 2020 Nov 11. PMID 33175656
- [Derived] Trimble CL, Morrow MP, Kraynyak KA, Shen X, Dallas M, Yan J, Edwards L, Parker RL, Denny L, Giffear M, Brown AS, Marcozzi-Pierce K, Shah D, Slager AM, Sylvester AJ, Khan A, Broderick KE, Juba RJ, Herring TA, Boyer J, Lee J, Sardesai NY, Weiner DB, Bagarazzi ML. Safety, efficacy, and immunogenicity of VGX-3100, a therapeutic synthetic DNA vaccine targeting human papillomavirus 16 and 18 E6 and E7 proteins for cervical intraepithelial neoplasia 2/3: a randomised, double-blind, placebo-controlled phase 2b trial. Lancet. 2015 Nov 21;386(10008):2078-2088. doi: 10.1016/S0140-6736(15)00239-1. Epub 2015 Sep 17. PMID 26386540